CLINICAL TRIAL: NCT05465746
Title: Correlation Between 24-hour Blood Pressure Load and Left Ventricular Mass: the CAPAMAVI
Brief Title: Cumulative Blood Pressure Load and Left Ventricular Mass
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Ecuatoriano del Corazón (Other)
Responsible Party: Sponsor
Other Study IDs: IECOR002
Record Dates: First submitted 2022-07-16; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Arterial Hypertension
Keywords: Ambulatory blood pressure monitoring; Blood pressure; Target organ damage; Left ventricular mass; Transthoracic echocardiography
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with an indication of SAH screening: Patients who attend the physician's office or the emergency room (ER) with signs and symptoms of high systemic arterial blood pressure will be indicated for ABPM and TTE
  Interventions: Diagnostic Test: 24-hour ambulatory blood pressure monitoring (ABPM); Diagnostic Test: Three-dimensional transthoracic echocardiography

INTERVENTIONS:
Diagnostic Test: 24-hour ambulatory blood pressure monitoring (ABPM) — Using a WatchBPO3 AFIB device (Microlife) placed around the left upper arm, BP measurements will be recorded every twenty minutes during the day and every thirty minutes at night, over a twenty-four-hour period. The device will automatically calculate the BP and the twenty-four-hour average BP, day, night, and cumulative BP load
Diagnostic Test: Three-dimensional transthoracic echocardiography — Using an EPIQ CVx (Philips) echocardiograph with an ultrasound sector transducer, 3D-TTE will be performed to assess the LVM index.

SUMMARY:
Delay in the diagnosis of systemic arterial hypertension (SAH) causes morbid hypertensive status with target organ damage (TOD). Screening and surveillance of SAH used to be performed through self-measurement of blood pressure (SMBP) or routinary in clinic blood pressure measurement (CBPM).

It is essential to determine the correlation between the cumulative blood pressure load through ABPM and the left ventricular mass identified by three-dimensional transthoracic ultrasound (3D-TTE). We postulate a directly proportional and statistically significant association between cumulative blood pressure load and left ventricular mass (LVM).

DETAILED DESCRIPTION:
Delayed diagnosis of SAH causes a morbid hypertensive state, with target-organ damage (TOD): brain, kidney, and heart. An early diagnosis and proper follow-up of patients with SAH prevents and reduces comorbidities associated with TOD. Screening and follow-up of SAH are traditionally performed by routine self-monitoring of blood pressure (HBPM) or clinic blood pressure measurement (CBPM).

Ambulatory blood pressure monitoring (ABPM) consists of measuring BP every fifteen and thirty minutes for twenty-four hours, using a sphygmomanometer adapted to a portable monitor, which led to the recognition of SAH phenotypes often not identified through SMBP or CBPM. The ABPM offers three types of information: a) the mean BP in twenty-four hours, day and night; b) BP variability; and c) cumulative BP load. Cumulative BP load is the percentage of BP measurements above 135/85 mmHg.

Increased LVM is a consequence of chronic hypertension and early sign of TOD at the cardiac level. It has been shown that the variability in nocturnal diastolic BP correlates significantly with LVM, independently of mean BP load. It is likely that an elevated BP load according to ABPM correlates with higher TOB; however, at the moment, there is no standardized value of BP load that allows predicting the increase in the LVM. For this reason, a standardized cut-off of cumulative BP load is helpful for understanding ABPM in the screening SAH.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Between 40 and 79 years old.
* Low or moderate cardiovascular risk according to the 3American Heart Association (AHA) criteria.

Exclusion Criteria:

* Patients with TOD defined as: the history of cerebrovascular event (CVD); chronic kidney disease (CKD) with glomerular filtration rate (GFR) <30 mL/min/1.73 m2 or under replacement therapy (renal dialysis).
* History of chronic liver disease with a Child-Pugh B or C.
* Dependence on alcohol or psychotropic drugs.
* History of cancer, regardless of stage or time of treatment.
* Patients who do not wish to participate in this study.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with an indication of SAH screening.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
24-hour systolic and diastolic blood pressure (SBP & DBP) | 24 hours
  The ABPM study will allow obtaining results of the mean BP in 24 hours, day and night; BP variability; and the pressure load. According to the international HBP guideline, normal BP will be considered below 135/85 mmHg during the twenty-four hours or during the day or below 120/70 mmHg at night. BP load is the percentage of BP measurements above 135/85 mmHg.
Left ventricular mass index (LVMI) | 30 minutes
  LVMI will be considered high when it exceeds 115 g/m2 of the body surface in men and 95 g/m2 in women. Each 3D-TTE will be performed by an echocardiographic cardiologist with experience in more than 5,000 3D-TTEs performed on adults annually. For the LVMI estimate to be as unbiased as possible, she will perform the 3D-TTE blind to any clinical history before completing the ABPM.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Delgado-Cedeño, MD, Principal Investigator — Instituto Ecuatoriano del Corazón
Locations (1):
- Instituto Ecuatoriano del Corazón, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cuspidi C, Sala C, Casati A, Bombelli M, Grassi G, Mancia G. Clinical and prognostic value of hypertensive cardiac damage in the PAMELA Study. Hypertens Res. 2017 Apr;40(4):329-335. doi: 10.1038/hr.2016.153. Epub 2016 Nov 17. PMID 27853165
- [Result] Mustafa ER, Istratoaie O, Musetescu R. Blood Pressure Variability and Left Ventricular Mass in Hypertensive Patients. Curr Health Sci J. 2016 Jan-Mar;42(1):47-50. doi: 10.12865/CHSJ.42.01.07. Epub 2016 Mar 29. PMID 30568812
- [Result] O'Brien E, White WB, Parati G, Dolan E. Ambulatory blood pressure monitoring in the 21st century. J Clin Hypertens (Greenwich). 2018 Jul;20(7):1108-1111. doi: 10.1111/jch.13275. PMID 30003702
- [Result] Uallachain GN, Murphy G, Avalos G. The RAMBLER study: the role of ambulatory blood pressure measurement in routine clinical practice: a cross-sectional study. Ir Med J. 2006 Oct;99(9):276-9. PMID 17144238
- [Result] Jones NR, McCormack T, Constanti M, McManus RJ. Diagnosis and management of hypertension in adults: NICE guideline update 2019. Br J Gen Pract. 2020 Jan 30;70(691):90-91. doi: 10.3399/bjgp20X708053. Print 2020 Feb. No abstract available. PMID 32001477